CLINICAL TRIAL: NCT02165410
Title: MRI Study of Cerebral Blood Flow in Development Disorders in Children
Acronym: IRM-Aut
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P120204; 2012-A01695-38 (Other: ANSM)
Record Dates: First submitted 2014-01-20; First posted 2014-06-17 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Autism
Keywords: Autism, mental retardation, Magnetic Resonance Imaging
MeSH Terms: conditions — Autistic Disorder; Intellectual Disability | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eye tracking and RMI (Experimental)
  Interventions: Procedure: ASL-MRI; Procedure: Diffusion tensor imaging (diffusion MRI); Procedure: Resting state MRI; Procedure: Eye-tracking; Procedure: Cognitive profile

INTERVENTIONS:
Procedure: ASL-MRI — ASL MRI is a non-invasive technique without injection to measure rCBF at rest marking the intravascular water molecules and use it as an endogenous tracer. Premedication, if required, will concern autistic and mentally retarded subjects only.
Procedure: Diffusion tensor imaging (diffusion MRI) — Diffusion MRI enables the mapping of the diffusion process of water molecules, which allows visualizing anatomical connections between different parts of the brain, noninvasively and on an individual basis. The sequence is acquired following clinical MRI sequences, while the child is still inside the MRI machine, with no further intervention applied.
Procedure: Resting state MRI — This sequence is based on the synchronization of fluctuations in the blood-oxygen level dependent (BOLD) signal of different brain regions that work as a network. Therefore this sequence allows for the establishing of maps of funcitonal connectivity.
Procedure: Eye-tracking — Eye tracking is a non-invasive method that allows objectifying gaze parameters during presentation of stimuli on a computer screen. Children will be presented with a series of social and no social stimuli and are required to watch it, with no further intervention applied.
Procedure: Cognitive profile — Children will be asked to perform certain tasks, adapted for their age.

SUMMARY:
The purpose of this study is reproduce the individual detection results by PET with Arterial Spin Labeling (ASL) MRI, to establish a biomarker useful in autism diagnosis.

DETAILED DESCRIPTION:
Anatomical and functional abnormalities have been identified in the superior temporal sulcus (STS) in autism by brain imaging modalities, including positron emission tomography (PET), functional MRI and diffusion MRI. These results suggest that brain imaging abnormalities within the STS could be the first step in the cascade of neuronal abnormalities found in autism.

STS is known as a key area for social cognition and is involved in various stages of social interaction, from visual and auditory perception (perception of eyes, facial and body movements, and perception of human voice) to the more complex process of social cognition (theory of mind, understanding emotions and mentalizing) The anatomical and functional abnormalities within the STS described in autism could account for the social difficulties experienced by persons with autism, both clinically observed and objectified by studies on visual social perception.

The individual detection results found in PET, that is to say a reduction of rCBF in the superior temporal sulcus (STS), could be reproduced with ASL and used to predict the diagnosis of autism in children with the same level of sensitivity and specificity as with PET. The individual detection of decreased rCBF in the STS could be a useful biomarker in autism using MRI, a method more accessible and much less invasive than PET. A MRI biomarker in autism could allow individual analysis, as well as contribute to early diagnosis and objective evaluation of the efficacy of new therapeutic strategies.

The rCBF data measured by MRI-ASL will also be correlated with both clinical (Autism Diagnostic Interview - ADI-R) and behavioral data of the social perception measured by the eye-tracking method. In addition, we will study the impact of these temporal anomalies on brain connectivity MRI method of diffusion tensor. We will also describe the abnormalities present in the very early development of autism.

ELIGIBILITY:
Inclusion Criteria:

Patient diagnosed autist or suspected autist : males and females with the diagnosis of autism based on the following criteria:

* 5 years ≤ age < 18 years,
* demand for MRI in the etiologic assessment (suspected autism) or MRI control in the treatment (diagnosed with autism)
* obtaining written consent from parents or legal guardians of patients.

Patients diagnosed with mental retardation or suspected with mental retardation : males and females with the diagnosis of mental retardation using the following criteria:

* 5 years ≤ age < 18 years,
* demand for MRI in the etiologic assessment (suspected mental retardation) or MRI control in the treatment (diagnosed with mental retardation)
* obtaining written consent from parents or legal guardians of patients.

Healthy control subjects: males and females:

* 5 years ≤ age < 18 years
* no known neurological or psychiatric disorder obtaining written consent with parents or legal guardians of volunteers.

Very young patients suspected of autism: male and female with suspected autism

1. 18 months ≤ age <5 years
2. demand of MRI in the etiologic assessment
3. obtaining written consent from parents or legal guardians.

Very young patients suspected of mental retardation : male and female with suspected mental retardation

1. 18 months ≤ age <5 years
2. demand of MRI in the etiologic assessment
3. obtaining written consent from parents or legal guardians.

All subjects must be registered with the social security.

Exclusion Criteria:

For all subjects:

* Indication against performing MRI (pacemaker, an implanted metal foreign body, claustrophobia),
* Inability of healthy volunteers to remain still during the MRI examination.

Healthy control subjects: males and females:

* aged between 5 years and 18 years
* no known neurological or psychiatric disorder
* obtaining written consent with parents or legal guardians of volunteers.

All subjects must be registered with the social security.

Exclusion Criteria:

For all subjects:

* Indication against performing MRI (pacemaker, an implanted metal foreign body, claustrophobia),
* Inability of healthy volunteers to remain still during the MRI examination.

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 175 (Estimated)
Dates: Start 2013-11-13 (Actual); Primary Completion 2023-09-13 (Estimated); Study Completion 2023-09-13 (Estimated)

PRIMARY OUTCOMES:
CBF | at day 0
  ASL is an MRI technique to measure CBF at rest by labeling arterial intravascular water and use as an endogenous tracer. This sequence is performed without injection of contrast or injection of radioactivity

SECONDARY OUTCOMES:
anatomical connectivity | at Day 0
  Diffusion tensor MRI (DTI) enables the mapping of the diffusion process of water molecules, which allows visualizing anatomical connections between different parts of the brain, noninvasively and on an individual basis.
eye-tracking method | at day 0
  Eye tracking is a non-invasive method that allows objectifying gaze parameters during presentation of stimuli on a computer screen.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie BODDAERT, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades Service de Radiologie Pédiatrique, Paris, France